CLINICAL TRIAL: NCT00492999
Title: A Phase II Study of the Rate of Conversion to Complete Resection in Patients With Initially Inoperable Hepatic-Only Metastases From Colorectal Cancer After Treatment With Hepatic Arterial Infusion With Floxuridine and Dexamethasone in Combination With Best Systemic Chemotherapy
Brief Title: Hepatic Arterial Infusion With Floxuridine and Dexamethasone Combined With Combination Chemotherapy in Treating Patients With Colorectal Cancer That Has Spread to the Liver
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-075; MSKCC-06075
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: recurrent colon cancer; stage IV colon cancer; recurrent rectal cancer; stage IV rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum; liver metastases
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — Dexamethasone; Floxuridine; Fluorouracil; Irinotecan; Leucovorin; Oxaliplatin

ARMS (2):
- Group 1 (Experimental): Patients receive hepatic arterial infusion (HAI) therapy comprising floxuridine and dexamethasone continuously on days 1-14. Patients also receive oxaliplatin IV over 2 hours and irinotecan hydrochloride IV over 30 minutes on days 1 and 15. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: dexamethasone; Drug: floxuridine; Drug: irinotecan hydrochloride; Drug: oxaliplatin
- Group 2 (Experimental): Patients receive HAI therapy as in group 1. Patients also receive irinotecan hydrochloride IV over 30 minutes and leucovorin calcium IV over 30 minutes on days 1 and 15 and fluorouracil IV continuously over 48 hours on days 1, 2, 15, and 16. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: dexamethasone; Drug: floxuridine; Drug: fluorouracil; Drug: irinotecan hydrochloride; Drug: leucovorin calcium

INTERVENTIONS:
Drug: dexamethasone — Given by hepatic arterial infusion
Drug: floxuridine — Given by hepatic arterial infusion
Drug: fluorouracil — Given IV
  Arms: Group 2
Drug: irinotecan hydrochloride — Given IV
Drug: leucovorin calcium — Given IV
  Arms: Group 2
Drug: oxaliplatin — Given IV
  Arms: Group 1

SUMMARY:
RATIONALE: Hepatic arterial infusion uses a catheter to carry tumor-killing substances directly into the liver. Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving floxuridine and dexamethasone directly into the arteries around the tumor together with combination chemotherapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well hepatic arterial infusion with floxuridine and dexamethasone works when given together with combination chemotherapy in treating patients with colorectal cancer that has spread to the liver.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the rate of conversion to complete resection in patients with initially unresectable colorectal cancer metastatic to the liver treated with hepatic arterial infusion comprising floxuridine and dexamethasone in combination with systemic irinotecan hydrochloride and either oxaliplatin or leucovorin calcium/fluorouracil.

Secondary

* Evaluate the time to progression in patients treated with this regimen.
* Evaluate disease-free survival of patients treated with this regimen.
* Evaluate overall survival of patients treated with this regimen.
* Determine the response rate (complete, partial, and moderate response) in patients treated with this regimen.
* Evaluate the safety profile and tolerability of this regimen in these patients.
* Assess the expression pattern of the VEGF receptor VEGFR1, VEGFR2, and VEGFR3 and their cognate ligands (i.e., VEGF-A, VEGF-B, VEGF-C, VEGF-D, and P1GF) in patients treated with this regimen.
* Correlate circulating angiogenic markers with tumor resectability, disease progression, and patient survival.
* Procure normal and diseased liver tissue for evaluation of thymidylate synthase, p53 gene, p21, topoisomerase 1, dihydropyrimidine dehydrogenase, and excision repair cross-complementing gene levels.
* Assess the expression pattern of tissue factor (TF) and explore its correlation with the TF receptors PAR-1, PAR-2, TF regulators PTEN, k-ras, b- raf, p53, and outcome.(Closed as of 11/30/10)
* Assess the prognostic and predictive role of preoperative, pretreatment, and during treatment serum TF in regards to outcome (progression-free survival and overall survival) and response to treatment with this regimen and to salvage treatments such as EGFR-inhibitors.(Closed as of 11/30/10)

OUTLINE: This is an open-label, nonrandomized study. Patients are assigned to 1 of 2 treatment groups according to receipt of more than 2 prior courses of oxaliplatin (no vs yes).

* Group 1 (no more than 2 prior courses of oxaliplatin): Patients receive hepatic arterial infusion (HAI) therapy comprising floxuridine and dexamethasone continuously on days 1-14. Patients also receive oxaliplatin IV over 2 hours and irinotecan hydrochloride IV over 30 minutes on days 1 and 15. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
* Group 2 (more than 2 prior courses of oxaliplatin): Patients receive HAI therapy as in group 1. Patients also receive irinotecan hydrochloride IV over 30 minutes and leucovorin calcium IV over 30 minutes on days 1 and 15 and fluorouracil IV continuously over 48 hours on days 1, 2, 15, and 16. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

In both groups, patients may undergo complete resection of liver metastases after completion of at least 3 courses of therapy.

Some patients undergo blood and tissue collection periodically for correlative and immunological studies. Samples are analyzed for VEGF receptor VEGFR1, VEGFR2, VEGFR3, thymidylate synthase, p53, p21, topoisomerase 1, dihydropyrimidine dehydrogenase, and excision repair cross-complementing gene levels.

After completion of study treatment, patients are followed every 3 months for 2 years, every 4 months for 3 years, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed colorectal adenocarcinoma metastatic to the liver

  * Previously treated or untreated disease
  * No clinical or radiographic evidence of extrahepatic disease
* Primary tumor may be present at study registration provided it is not obstructing the intestinal lumen or is significantly bleeding

  * If present, the primary tumor will be resected at the time of pump placement
* Must have inoperable liver metastases confirmed by 2-3 hepatobiliary surgeons and the assigned radiologist

  * Liver metastases < 70% of the liver parenchyma
  * Inoperable liver metastases is defined by one of the following:

    * More than 6 metastases in a single lobe with one lesion ≥ 5 cm
    * At least 6 metastases distributed diffusely in both lobes of the liver
    * When a margin-negative resection would require resection of all three hepatic veins, both portal veins, or the retrohepatic vena cava
    * Requires a resection that leaves < 2 hepatic segments (not including the caudate lobe) behind with adequate arterial or portal inflow, venous outflow, and biliary drainage
* No ascites or hepatic encephalopathy
* No history of primary CNS tumors

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* WBC ≥ 3,000/mm^3
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* INR < 1.5
* Hemoglobin ≥ 9 g/dL
* Creatinine ≤ 1.5 mg/dL
* Total bilirubin ≤ 1.5 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Physically able to tolerate major partial hepatectomy
* No active infection
* No concurrent active malignancies, except potentially resectable primary colorectal tumor
* No bleeding diathesis or coagulopathy
* No history of serious systemic disease, including any of the following:

  * Myocardial infarction within the past 6 months
  * Uncontrolled hypertension (i.e., blood pressure > 150/100 mm Hg on medication)
  * Unstable angina
  * New York Heart Association class II-IV congestive heart failure
  * Unstable symptomatic arrhythmia requiring medication

    * Chronic atrial arrhythmia (i.e., atrial fibrillation or paroxysmal supraventricular tachycardia) allowed
  * Peripheral vascular disease ≥ grade 2
* No serious or nonhealing active wound, ulcer, or bone fracture
* No history of seizures not well controlled with standard medical therapy
* No stroke or transient ischemic attack within the past 6 months
* No concurrent obstruction of the gastrointestinal or genitourinary tract

PRIOR CONCURRENT THERAPY:

* At least 4 weeks since prior radiotherapy to the pelvis
* Prior chemotherapy allowed
* No prior radiotherapy, hepatic thermal ablation, or resection (other than biopsy) to the liver
* No prior floxuridine
* No prior hepatic arterial infusion
* No concurrent chronic aspirin (> 325 mg/day) or nonsteroidal anti-inflammatory medications known to inhibit platelet function
* No other concurrent investigational agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2007-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Resectability rate | 2 years

SECONDARY OUTCOMES:
Antitumor activity | 2 years
Response rate | 2 years
Median time to progression | 2 years
Survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael D'Angelica, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Nancy E. Kemeny, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York
  - Memorial Sloan Kettering Cancer Center@Phelps Memorial Hospital, Sleepy Hollow, New York

REFERENCES:
- [Derived] Correa-Gallego C, Gavane S, Grewal R, Cercek A, Klimstra DS, Gewirtz AN, Kingham TP, Fong Y, DeMatteo RP, Allen PJ, Jarnagin WR, Kemeny N, D'Angelica MI. Prospective evaluation of 18F-fluorodeoxyglucose positron emission tomography in patients receiving hepatic arterial and systemic chemotherapy for unresectable colorectal liver metastases. HPB (Oxford). 2015 Jul;17(7):644-50. doi: 10.1111/hpb.12421. Epub 2015 May 23. PMID 26010778
- [Derived] D'Angelica MI, Correa-Gallego C, Paty PB, Cercek A, Gewirtz AN, Chou JF, Capanu M, Kingham TP, Fong Y, DeMatteo RP, Allen PJ, Jarnagin WR, Kemeny N. Phase II trial of hepatic artery infusional and systemic chemotherapy for patients with unresectable hepatic metastases from colorectal cancer: conversion to resection and long-term outcomes. Ann Surg. 2015 Feb;261(2):353-60. doi: 10.1097/SLA.0000000000000614. PMID 24646562
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm